CLINICAL TRIAL: NCT05481996
Title: Effectiveness of an Exercise-based Telerehabilitation Program for Police Officers and Firefighters With Chronic Non-specific Low Back Pain: a Randomized Clinical Trial
Brief Title: Exercise-based Telerehabilitation Program for Police Officers and Firefighters With Chronic Non-specific Low Back Pain
Acronym: SAFEBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Cristine Lima Alberton, PhD, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 58715422.3.0000.5313
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Chronic Low-back Pain; Telerehabilitation
Keywords: low back pain; Telerehabilitation
MeSH Terms: conditions — Low Back Pain | interventions — Exercise; Telerehabilitation

STUDY DESIGN:
Intervention Model Description: The Intervention group will perform the 8-week treatment with access to 8 pain education messages (1 message/week) and 8 weeks of an exercise program prescribed for people with chronic low back pain, and the control group will receive information on chronic low back pain for one booklet and access to 8 pain education messages (1 message/week). Randomized through software, so that the subject enters his/her login and password and is directed to one of the study groups, with a blind evaluator without access to randomization information throughout the study and follow-up of the outcome measures for 4 months after randomization.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-Based Pain Education and Exercise (Experimental): Patients allocated to the experimental group will receive a login and password for individual access to the smartphone app designed for the study. The app's content for this group will include three components: 1) a physical exercise program of 8 weeks; 2) weekly messages; and 3) an online booklet. The exercise component will include 8 weeks of training, with two sessions per week of core strengthening exercises. The app will provide illustrations, with animated images (GIFs), descriptions and audios of how to perform each exercise. The message component will provide eight messages (one per week), which will have their contents taken from the online booklet. Messages will include information about the benefits of exercise, motivation, and positive messages about coping with pain. The online booklet will contain general information about self-management of chronic pain, including pain education, advice on healthy lifestyle and sleeping habits and promotion of exercises.
  Interventions: Other: App-Based Pain Education and Exercise
- Online Booklet (Active Comparator): Patients allocated to the control group will receive a login and password for individual access to the smartphone app designed for the study. The app's content for this group will include two components: 1) an online booklet; and 2) weekly messages. The online booklet will contain general information about self-management of chronic pain, including pain education, advice on healthy lifestyle and sleeping habits and promotion of exercises. The message component will provide eight messages (one per week), which will have their contents taken from the online booklet. Messages will include information about the benefits of exercise, motivation, and positive messages about coping with pain.
  Interventions: Other: Online booklet

INTERVENTIONS:
Other: App-Based Pain Education and Exercise — Telerehabilitation is defined as providing techniques for therapeutic rehabilitation remotely or off-site using telecommunication technologies. Thus, our intervention will be based on the use of a smartphone application created especially for the study that will contain a program of progressive physical exercises with images and descriptions, educational messages and an online booklet for the study subjects, totaling 8 weeks of training and pain education.
  Other Names: Telerehabilitation
  Arms: App-Based Pain Education and Exercise
Other: Online booklet — An online booklet containing information about chronic low back pain and weekly messages about low back pain causes, suggestions for lifestyle modifications and behavior will be delivered, as well as an incentive to perform physical exercises.
  Arms: Online Booklet

SUMMARY:
The aim of this clinical trial is to develop and test the effectiveness of a smartphone app-based self-management program based on exercise and pain education for police officers and firefighters with chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is the leading cause of year lived with disability worldwide. Workers exposed to physically demanding activities and inappropriate postures, such as those performed by police officers and firefighters, are highly affected by chronic low back pain. Smartphone app-based self-managed interventions have been shown to be an alternative for chronic non-specific low back pain treatment. However, there is still little research on the development and testing of remotely-delivered programs for the management of chronic low back pain, especially in police and fire professionals. The aim of this clinical trial is to develop and test the effectiveness of a smartphone app-based self-management program based on exercise and pain education for police officers and firefighters with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years
* Chronic low back pain (defined as pain lasting more than 12 weeks)
* Chronic low back pain of at least 3 points in a 0 to 10 Pain Numerical Rating Scale
* Own a smartphone with internet access and email account
* Police officer (federal, federal highway, civil or military) or military firefighter working in the State of Rio Grande do Sul

Exclusion Criteria:

* Present neurological symptoms (nerve root compromise, or sensation deficits)
* Present serious spinal diseases (e.g., fracture, tumor, inflammatory, autoimmune, and infectious diseases)
* Present serious cardiovascular and metabolic diseases (e.g., coronary heart disease, cardiac insufficiency, decompensated diabetes)
* Recent spine surgery (over the last 12 months) or scheduled to undergo surgery in the next six months, or pregnancy
* History of physical therapy treatment for low back pain or physical exercise (strength training for core muscles, Pilates, yoga) current or within the last 3 months
* Retired
* If have any contraindication to exercise:

We will perform a pre-screening for physical activity participation at baseline using the Physical Activity Readiness Questionnaire (PAR-Q) Portuguese version to rule out any contraindication to participate in physical activity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity at post-treatment follow-up | Post-treatment follow-up (8 weeks)
  The primary outcome will be pain intensity measured using the Pain Numerical Rating Scale, a numerical scale of 11 domains, where 0 indicates no pain and 10 indicates maximum pain intensity.
Disability at post-treatment follow-up | Post-treatment follow-up (8 weeks)
  The primary outcome will be disability measured using the Roland Morris Disability Questionnaire, a 24-item questionnaire that assesses normal activities of daily living, where a higher score indicating a higher level of disability.

SECONDARY OUTCOMES:
Pain intensity at 4 months follow-up | 4 months follow-up
  Measured using the Pain Numerical Rating Scale, a numerical scale of 11 domains, where 0 indicates no pain and 10 indicates maximum pain intensity.
Disability at 4 months follow-up | 4 months follow-up
  Measured using the Roland Morris Disability Questionnaire, a 24-item questionnaire that assesses normal activities of daily living, where a higher score indicating a higher level of disability.
Health-Related Quality of Life | The outcome will be evaluated after the treatment period (8 weeks) and after 4 months of randomization of each subject.
  Measured with the WHOQOL-Pain, a self-reported questionnaire with 16 questions and classification of 4 facets related to the experience of chronic physical pain.
Self-efficacy | The outcome will be evaluated after the treatment period (8 weeks) and after 4 months of randomization of each subject.
  Measured with Pain Self-Efficacy Questionnaire, a questionnaire with 22 questions classified in three domains, with a score of each domain ranging from 10 to 100. A total score close to 300 indicates a greater sense of self-efficacy.
Depression, Anxiety and Stress | The outcome will be evaluated after the treatment period (8 weeks) and after 4 months of randomization of each subject.
  Measured by the Depression Anxiety Stress Scale, a self-reported scale with 21 questions, 7 for depression, 7 for anxiety and 7 for stress. Each question ranges from 0 to 3 according to the patient's response. Scores near 21 indicate the worst results.
Sleep quality | The outcome will be evaluated after the treatment period (8 weeks) and after 4 months of randomization of each subject.
  Measured by the Pittsburgh Sleep Quality Index, a self-reported scale with 19 questions, that assess seven components of sleep. Each question ranges from 0 to 3 according to the patient's response. Scores near 21 indicate worse sleep quality.
Work ability | The outcome will be evaluated after the treatment period (8 weeks) and after 4 months of randomization of each subject.
  Measured by a single-item question: Are you working at a physically less demanding job now because of your back and/or leg pain?
Isometric muscular endurance of the trunk extensor | The outcome will be evaluated after the treatment period (8 weeks).
  Measured by modified Biering-Sorensen test.
Isometric muscular endurance of the trunk flexors | The outcome will be evaluated after the treatment period (8 weeks).
  Measured by a test that consists of remaining in isometry as long as possible.
Maximum isometric strength of the trunk extensor and flexor muscles | The outcome will be evaluated after the treatment period (8 weeks).
  Measured by a load cell.
Muscular activation of flexor and extensor muscles | The outcome will be evaluated after the treatment period (8 weeks).
  Measured using the surface electromyography technique. The neuromuscular activation of flexor (rectus abdominis) and extensor (spinal erector) muscles will be measured.
Adverse Effects | The outcome will be evaluated after the treatment period (8 weeks) and after 4 months of randomization of each subject.
  Measured by recording the number of adverse events during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Cristine Alberton, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Escola Superior de Educação Física, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marins EF, Caputo EL, Kruger VL, Junior DM, Scaglioni FG, Del Vecchio FB, Primo TT, Alberton CL. Effectiveness of m-health-based core strengthening exercise and health education for public safety workers with chronic non-specific low back pain: study protocol for a superiority randomized controlled trial (SAFEBACK). Trials. 2023 Dec 1;24(1):780. doi: 10.1186/s13063-023-07833-9. PMID 38041180